CLINICAL TRIAL: NCT00767312
Title: Analysis of HIV-1 Replication During Antiretroviral Therapy
Status: Enrolling by invitation | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080221; 08-I-0221
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2025-09-24 (Actual); Status verified 2025-09-12

CONDITIONS: HIV
Keywords: HIV; Natural History

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: HIV-infected patients who are 18 years of age or older, have been enrolled in another NIH protocol.

SUMMARY:
This study will determine if the level of virus in HIV-infected patients taking antiretroviral medications for prolonged periods decreases or persists at a stable level. It will also examine whether new gene changes (mutations) occur during drug suppression.

HIV-infected patients who are 18 years of age or older, have been enrolled in another NIH protocol, have been suppressed on antiretroviral therapy and have very low levels of virus in their blood may be eligible for this 5-year (or more) study.

Participants come to the NIH Clinical Center about every 6 months for a physical examination, routine and research blood tests and leukapheresis to collect white blood cells for T cell analysis. For leukapheresis, blood is collected through a vein much like donating whole blood, but the blood is directed through a machine that separates and extracts the white cells and returns the rest of the blood components to the patient. Patients may also have an optional third clinic visit each year for another blood draw.

DETAILED DESCRIPTION:
Combination antiretroviral therapy for human immunodeficiency virus serotype 1 (HIV-1) infection has resulted in profound reductions in viremia and is associated with marked improvements in morbidity and mortality. Therapy is not curative, however, and prolonged therapy is complicated by drug toxicity and the emergence of drug resistance. How drug resistance emerges during suppressive antiretroviral therapy remains poorly understood. Investigating the characteristics of HIV-1 replication during suppressive antiretroviral therapy will yield important insights in understanding the emergence resistance, and requires patients who have suppressed viral RNA levels. Prior National Institutes of Health (NIH) protocols have made important observations regarding the kinetics of HIV-1 decline in response to therapy, the levels of HIV-1 viremia during suppressive therapy, and the nature of HIV-1 genetic diversity prior to and following initiation of antiretroviral therapy. In the process, these studies have generated a useful cohort of patients with suppressed viral RNA levels, who have been extensively characterized from a virologic and immunologic standpoint. Similarly, patients from other NIH protocols have been followed for prolonged periods before and after therapy has been initiated, and they also have stored sample sets that would be useful in new studies of HIV replication. The HIV Drug Resistance Program (DRP) has studied samples from protocols 00-I-0110 and 97-I-0082 to develop a number of new, sensitive laboratory techniques to measure and quantitate genetic variation and to investigate immune response parameters. To further advance understanding of HIV-1 replication during suppressive antiretroviral therapy and the emergence of drug resistance, we propose a new protocol to study these 2 patient cohorts (from the above cited protocols) and selected patients in other protocols with a new series of studies. The primary objective of this protocol is to investigate the virologic and immunologic characteristics of HIV-infected individuals undergoing antiretroviral therapy. Upon implementation, this new protocol will provide human subjects protection for samples collected under the two prior protocols, whether patients enroll in the new study or not.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion criteria for this protocol comprise all of the following conditions:

* Age greater than or equal to 18 years.
* HIV infection with documented reactive ELISA and positive western blot.
* Prior enrollment in 00-I-0110, 97-I-0082 OR patients with long term evaluation at NIH for whom additional sampling will be useful for protocol objectives, including:

  * Available stored specimens from pretherapy period.
  * Ongoing suppression of viremia with bDNA less than 50 copies/mL, OR
  * Suppression of viremia to less than 50 copies/mL followed by rebound viremia during therapy.
* Patients must have a private physician for routine medical care.

EXCLUSION CRITERIA:

Any prospective study subject who has been previously withdrawn from any prior study for inability to comply with study procedures will be considered ineligible for this study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from studies: 00-I-0110 and 97-I-0082 are eligible for enrollment. Patients in other NIH studies would be considered for co-enrollment in this study if continued longitudinal sample acquisition is deemed desirable.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2008-11-17 (Actual)

PRIMARY OUTCOMES:
We plan to investigate the relationship of HIV-1 viral RNA levels and genetic variation in patients on antiretroviral therapy over prolonged periods. | every 6 months
  HIV-1 viral RNA

SECONDARY OUTCOMES:
Provide human subjects protection oversight for samples accrued in protocol 97-I-0082 and 00-I-0110 | ongoing
  protection
Investigate the genetic and immunologic characteristics of patients with HIV-1 suppression on antiretroviral therapy who experience rebound viremia | ongoing
  genetic and immunologic
Investigate determinants of HIV-1 DNA quantity and characteristics in suppressed patients | ongoing
  HIV DNA quantity and characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Frank Maldarelli, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Identified data in BTRIS (automatic for activities in the Clinical Center).@@@@@@@@@@@@De-identified or identified data with approved outside collaborators under appropriate agreements.
Supporting Information: Study Protocol, ICF
Time Frame: Identified data in BTRIS (automatic for activities in the Clinical Center and will be available for use following the BTRIS Policy for Data Sharing and Use).
Access Criteria: Identified data in BTRIS (automatic for activities in the Clinical Center and will be available for use following the BTRIS Policy for Data Sharing and Use).@@@@@@@@@@@@De-identified or identified data with approved outside collaborators under appropriate agreements.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2008-I-0221.html